CLINICAL TRIAL: NCT00856713
Title: A Study in Healthy Volunteers and Patients With Liver Cirrhosis to Assess the Effects of Age, Gender, and Stable Liver Disease on the Clearance of Cholyl-Lysyl-Fluorescein (NRL972) as an in-Vivo Marker of Liver Function in Man
Brief Title: Clearance of NRL972 in Patients With Cirrhosis and in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President Clinical Development, Norgine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL972-01/2005 (ACPS)
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Hepatic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — NRL972

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 YM (Experimental): Healthy young males
  Interventions: Drug: NRL972
- 2 EM (Experimental): Healthy elderly males
  Interventions: Drug: NRL972
- 3 YF (Experimental): Healthy young females
  Interventions: Drug: NRL972
- 4 EF (Experimental): Healthy elderly females
  Interventions: Drug: NRL972
- 5 CTP-A (Experimental): Patients with hepatic cirrhosis CTP-class A
  Interventions: Drug: NRL972
- 6 CTP-BC (Experimental): Patients with hepatic cirrhosis CTP-class B and C
  Interventions: Drug: NRL972

INTERVENTIONS:
Drug: NRL972 — Single intravenous dose of 2 mg NRL972
  Arms: 1 YM
Drug: NRL972 — Single intravenous dose of 2 mg NRL972
  Arms: 2 EM
Drug: NRL972 — Single intravenous dose of 2 mg NRL972
  Arms: 3 YF
Drug: NRL972 — Single intravenous dose of 2 mg NRL972
  Arms: 4 EF
Drug: NRL972 — Single intravenous dose of 2 mg NRL972
  Arms: 5 CTP-A
Drug: NRL972 — Single intravenous dose of 2 mg NRL972
  Arms: 6 CTP-BC

SUMMARY:
A study in healthy volunteers and patients with liver cirrhosis to assess the effects of age, gender, and stable liver disease on the clearance of cholyl-lysyl-fluorescein (NRL972)

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following conditions will be eligible for enrolment:

General - all subjects

1. Males or females (females of non-child-bearing potential or of child-bearing potential while taking medically appropriate contraception)
2. Caucasian
3. BMI: between 19 and 34 kg.m-2
4. BW: between 45 and 110 kg
5. willing and able to provide informed consent

   Healthy volunteers (group N)
6. Age: 18 - 40 years (inclusive) and > 60 years
7. Assessed as healthy based on the pre-study examination

   Hepatic cirrhosis
8. Age: 18 - 75 years
9. stable compensated liver cirrhosis (cryptogenic, posthepatic, alcoholic) with histo-logical or macroscopic (e.g. laparascopy, biopsy, ultrasound sonography or other adequate imaging techniques) confirmation

Exclusion Criteria:

Subjects of any of the following categories will be excluded from enrolment:

General - all subjects

1. Previous participation in the trial
2. Participant in any other trial during the last 90 days
3. Donation of blood during the last 60 days or a history of blood loss exceeding 300 mL within the last 3 months
4. History of any clinically relevant allergy
5. Presence of acute or chronic infection
6. Uncontrolled diabetes mellitus
7. Resting systolic blood pressure > 160 or < 90 mmHg, diastolic blood pressure > 95 or < 50 mmHg
8. Clinically relevant ECG-abnormalities, prolonged QTc with > 450 msec in males and > 460 msec in females in particular
9. Positive HIV test
10. Positive alcohol or urine drug test on recruitment
11. Daily use of > 30 gr alcohol
12. Smoking more than 15 cigarettes/day or equivalent of other tobacco products
13. Use of prohibited medication
14. Suspicion or evidence that the subject is not trustworthy and reliable
15. Suspicion or evidence that the subject is not able to make a free consent or to under-stand the information in this regard

    General - all females
16. Positive pregnancy test
17. Lactating
18. Not using appropriate contraception in premenopausal women

    All healthy subjects
19. Presence or history of any relevant comorbidity
20. Presence of any relevant abnormality in the laboratory safety tests, especially low Hemoglobin, increased liver enzymes, reduced serum creatinine
21. Positive serology for HBsAg, anti HBc and anti HCV
22. History of alcohol and/or drug abuse

    Patients with hepatic disease
23. Biliary liver cirrhosis
24. Liver impairment due to space-occupying processes (e.g. carcinoma)
25. State after liver transplantation or patient scheduled for liver transplantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2006-03; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Clearance of NRL972 in healthy subjects and patients with hepatic cirrhosis | Up to 4 hrs post administration of NRL972

SECONDARY OUTCOMES:
Adverse events and changes in physical findings from baseline | Up to 4 hours post-dosing
Effects on vital signs: blood pressure, pulse rate | Up to 4 hours post-dosing
Effects on electrocardiogram | Up to 4 hours post-dosing
Changes in haematology, clinical chemistry, urinalysis | Up to 4 hours post-dosing

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine; Zahariy Krastev, MD, Principal Investigator — St Ivan Rilski's University Hospital
Locations (1):
- UMHAPT St Ivan Rilski's University Hospital, Sofia, Bulgaria